CLINICAL TRIAL: NCT02807909
Title: An Open-Label Single-Sequence Study to Evaluate the Effect of Co-administration of Itraconazole or Diltiazem on the Single-Dose Pharmacokinetics of BMS-986177 in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Co-administration of Itraconazole or Diltiazem on the Pharmacokinetics of BMS-986177 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV010-005
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-986177 and Itraconazole (Experimental): Single dose BMS-986177 on day 1 followed by Itraconazole and BMS-986177 on specified days
  Interventions: Drug: BMS-986177; Drug: Itraconazole
- BMS-986177 and Diltiazem (Experimental): Single dose BMS-986177 on day 1 followed by Diltiazem ER and BMS-986177 on specified days
  Interventions: Drug: BMS-986177; Drug: Diltiazem ER

INTERVENTIONS:
Drug: BMS-986177
Drug: Itraconazole
  Arms: BMS-986177 and Itraconazole
Drug: Diltiazem ER
  Arms: BMS-986177 and Diltiazem

SUMMARY:
The study is being conducted to assess the effects of co-administration of itraconazole or diltiazem, respectively, on the pharmacokinetic (PK) parameters Cmax, AUC(INF), and AUC(0-T) of BMS-986177

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy subjects as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory determinations.
3. Subjects with body mass index of 18 to 30 kg/m2, inclusive
4. Men, and women of nonchildbearing potential. Women must have documented proof that they are not of childbearing potential and are not breast feeding
5. Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of the study drug (3 days) plus 90 days (duration of sperm turnover) for a total of 92 days for subjects in the BMS-986177 - diltiazem sequence, and 99 days for subjects in the BMS-986177 - itraconazole sequence.

Exclusion Criteria:

1. Any significant acute or chronic medical illness, including hepatic disease, or any other condition listed as a contraindication in the diltiazem or itraconazole package inserts.
2. Evidence of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising or thrombus formation.
3. History of chronic constipation, GI disease, arrhythmias, sinus bradycardia, significant head injury, dizziness or headaches, hemophilia, Rosenthal syndrome, or FX1a deficiency or other coagulopathies, systemic lupus erythematosus.
4. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
5. History of allergy to BMS-986177, itraconazole, diltiazem, or related compounds.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC (0-T)) of BMS-986177 | Days 1-12
Maximum observed concentration (Cmax) | Days 1-12
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Days 1-12

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Screening- until 30 days after discontinuation of dosing or subject's participation in the study if the last scheduled visit occurs at a later time.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Perera V, Wang Z, Lubin S, Christopher LJ, Chen W, Xu S, Seiffert D, DeSouza M, Murthy B. Effects of Itraconazole and Diltiazem on the Pharmacokinetics and Pharmacodynamics of Milvexian, A Factor XIa Inhibitor. Cardiol Ther. 2022 Sep;11(3):407-419. doi: 10.1007/s40119-022-00266-6. Epub 2022 May 31. PMID 35641780
- See also: Description BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Description FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Description Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx